CLINICAL TRIAL: NCT05258773
Title: A Phase IIa, Multicenter, Randomized, Controlled, Open-label Study to Evaluate the Presence of SENS-401 in the Perilymph After 7 Days of Repeated Oral Administration in Adult Participants Scheduled for Cochlear Implantation
Brief Title: Evaluation of the Presence of SENS-401 in the Perilymph
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sensorion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SENS-401-203; 2021-006615-28 (EudraCT Number)
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — SENS-401

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- A, Treatment arm (Experimental): Arm A: Participants scheduled for cochlear implantation and treated with oral 43.5 mg SENS-401 (R-Azasetron Besylate) twice daily for up to 49 days.
  Interventions: Drug: SENS-401 (R-Azasetron Besylate)
- B, Control arm (No Intervention): Arm B: Participants scheduled for cochlear implantation and not treated with SENS-401 (R-Azasetron Besylate).

INTERVENTIONS:
Drug: SENS-401 (R-Azasetron Besylate) — Patients will receive SENS-401 ((R)-azasetron besylate) for 7 days B.I.D. before cochlear implant surgery and during 6 weeks after the surgery.
  Arms: A, Treatment arm

SUMMARY:
The aim of this study is to detect the presence of SENS-401 in the perilymph of participants undergoing cochlear implant surgery after 7 days of oral administration of SENS-401.

DETAILED DESCRIPTION:
The study is a Phase IIa, open-label, randomized and controlled study investigating repeated twice-daily administration of oral SENS-401 in adult participants with moderately severe to profound hearing loss who have already agreed to undergo cochlear implant surgery justified by their hearing impairment.

After written informed consent is obtained and screening procedures completed, 27 eligible participants will be randomized on Day 1 to either Arm A or Arm B in ratio 2:1 (18 participants in Arm A and 9 participants in Arm B).

Arm A participants will commence dosing with twice-daily oral 43.5 mg SENS-401 for 7 days prior to their scheduled cochlear implant surgery on Day 8 and up to 42 days from day of surgery inclusive.

Arm B participants will not receive any treatment other than their scheduled cochlear implant surgery.

ELIGIBILITY:
Main Inclusion Criteria:

Potential participants must fulfil all of the following main inclusion criteria to be eligible for the study:

1. Adults aged from 18 years and older;
2. Meets the locally approved indication for cochlear implantation. The individual must have freely consented to the cochlear implant surgery before being offered to participate in the SENS-401-203 study;
3. Signed and dated written informed consent;

Main Exclusion Criteria:

Individuals will be excluded from the study if any of the following main exclusion criteria apply:

1. Moderate to severe renal impairment defined by a creatinine clearance ≤ 60 ml/min
2. Any condition that, in the opinion of the Investigator, may compromise the safety or compliance of the participant or would preclude the participant from successful completion of the study
3. Unable or unwilling to comply with the protocol requirements
4. Known hypersensitivity, allergy or intolerance to the study medication or any history of severe abnormal drug reaction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen O'Leary, MD, Principal Investigator — Royal Victoria Eye and Ear Hospital
Locations (7):
- Royal Victorian Eye and Ear Hospital, Melbourne, Australia
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux, Hôpital Pellegrin, Bordeaux
  - Centre Hospitalier Universitaire de Clermont-Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Lille Hôpital Roger Salengro, Lille
  - Hôpital Edouard Herriot, Lyon
  - Groupe Hospitalier La Pitié-Salpétrière, Paris
  - Centre Hospitalier Universitaire de Toulouse, Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- B, Control Arm: Arm B: Participants scheduled for cochlear implants and not treated with SENS-401 (R-Azasetron Besylate).
Period: Overall Study
Arm/Group | A, Treatment Arm | B, Control Arm
Started | 18 | 10
Completed | 16 | 8
Not Completed | 2 | 2
Not completed — Screen Failure | 1 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised of all randomized participant. One (1) participant randomized in Arm A was excluded from the FAS due to the failure to satisfy major entry criteria, failure to take at least one dose of SENS-401 and the lack of any data post randomization.
  Seventeen (17) participants who received at least one dose of SENS-401 and all 10 participants randomized to no treatment, were included in the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | A, Treatment Arm | B, Control Arm | Total
Number analyzed (Participants) | 17 | 10 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.67 (13.602) | 61.52 (14.968) | 61.61 (13.835)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 5 | 4 | 9
  France | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With SENS-401 Detected in Perilymph
Description: A sample of perilymph was obtained from the round window during the cochlear implant surgery from Arm A participants only, after seven days of SENS-401. The percentage of participants with levels of SENS-401 in the perilymph above the Limit of Quantification was then calculated.
Time Frame: Day 8
Population: The pharmacokinetic (PK) Set included all participants who received at least one dose of SENS-401 (16). Note that one (1) participant treated with SENS-401 did not have a perilymph sample collected during cochlear implant surgery so the overall number of participants analyzed for this outcome is 15.
Measure: Count of Participants; unit: Participants
Arm/Group | A, Treatment Arm | B, Control Arm
Number analyzed (Participants) | 15 | 0
Participants | 15 | 0

2. Secondary Outcome: SENS-401 Perilymph Concentration
Description: SENS-401 perilymph concentration on day of cochlear implant surgery after seven days of SENS-401 (arm A only).
Time Frame: Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | A, Treatment Arm | B, Control Arm
Number analyzed (Participants) | 15 | 0
ng/ml | 45.8009 (45.47158) |

3. Secondary Outcome: SENS-401 Plasma Concentration
Description: SENS-401 plasma concentration on day of cochlear implant surgery after seven days of SENS-401 (arm A only).
Time Frame: Day 8
Population: The pharmacokinetic (PK) Set included all participants who received at least one dose of SENS-401 (16).
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | A, Treatment Arm | B, Control Arm
Number analyzed (Participants) | 16 | 0
ng/ml | 59.6244 (27.98319) |

4. Secondary Outcome: Change of Hearing Threshold From Baseline in the Implanted Ear at Several Frequencies
Description: Pure tone audiometry (PTA) in decibels (dB) is a behavioral, subjective hearing test used to assess an individual's hearing threshold levels and determine the degree of hearing loss. A decrease of hearing threshold is considered as an improvement and an increase as a deterioration of the audition.
  PTA assessments were conducted on Day 1 after randomization (prior to the first dose of the study drug for Arm A), at the Day 49 visit, and at the end of the study (EOS) on Day 105 for all participants (Arms A and B).
  The change in hearing threshold from baseline in the implanted ear was evaluated at 500 Hz and as an average across three frequencies (250, 500, and 750 Hz) using PTA.
Time Frame: Day 49 and Day 105
Population: Efficacy Set included all participants who have at least hearing threshold parameter data at Baseline and Day 49
Measure: Least Squares Mean (95% Confidence Interval); unit: dB
Arm/Group | A, Treatment Arm | B, Control Arm
Number analyzed (Participants) | 16 | 8
dB
  Day 49 : LS Mean change from baseline at 500Hz | 19.7 [11.1 to 28.2] | 30.6 [18.5 to 42.8]
  Day 49 : LS Mean change from baseline at 250-750 Hz: number analyzed (Participants) | 15 | 7
  Day 49 : LS Mean change from baseline at 250-750 Hz | 16.25 [7.92 to 24.59] | 30.65 [18.42 to 42.88]
  Day 105: LS Mean change from baseline at 500 Hz | 25.6 [16.4 to 34.8] | 34.5 [21.5 to 47.6]
  Day 105: LS Mean change from baseline at 250-750 Hz: number analyzed (Participants) | 15 | 7
  Day 105: LS Mean change from baseline at 250-750 Hz | 20.97 [11.63 to 30.32] | 34.82 [21.10 to 48.53]
Statistical Analysis 1: Comparison: A, Treatment Arm vs B, Control Arm; Test type: Superiority; p = 0.1406, ANCOVA — An analysis of covariance (ANCOVA) model was used to assess changes from baseline at 500Hz at the Day 49 visit comparing the treatment groups.The treatment group was included as a fixed factor, with baseline values as a covariate; LS Mean difference Arm A - Arm B = -11.0, 95% CI 2-sided [-25.9 to 3.9] — The change in hearing threshold from baseline was expected to be smaller in the treated group (arm A) than in the control group (arm B)
Statistical Analysis 2: Comparison: A, Treatment Arm vs B, Control Arm; Test type: Superiority; p = 0.0567, ANCOVA — An ANCOVA model was used to assess changes from baseline at the average across three frequencies (250-750 Hz) at the Day 49 visit comparing the treatment groups. The treatment group was included as a fixed factor, with baseline values as a covariate; LS Mean difference Arm A - Arm B = -14.40, 95% CI 2-sided [-29.24 to 0.45] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: A, Treatment Arm vs B, Control Arm; Test type: Superiority; p = 0.2588, ANCOVA — An ANCOVA model was used to assess changes from baseline at 500Hz at EOS on Day 105 comparing the treatment groups.The treatment group was included as a fixed factor, with baseline values as a covariate; LS Mean difference Arm A - Arm B = -9.0, 95% CI 2-sided [-25.0 to 7.1] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: A, Treatment Arm vs B, Control Arm; Test type: Superiority; p = 0.0979, ANCOVA — An ANCOVA model was used to assess changes from baseline at the average across three frequencies (250-750 Hz) at EOS on Day 105, comparing the treatment groups. The treatment group was included as a fixed factor, with baseline values as a covariate; LS Mean difference Arm A - Arm B = -13.84, 95% CI 2-sided [-30.49 to 2.80] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: 105 days
Description: Adverse events were recorded for all study participants from the time of informed consent to study completion. For arm A other adverse events reported below areTreatment Emergent Adverse Events defined as follow: any untoward medical occurrence reported or observed after treatment administration.
  Safety assessments were performed at every site visit for all participants: regular investigator assessment and regular laboratory testing
Arm/Group | A, Treatment Arm | B, Control Arm
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/17 | 0/10
Other Adverse Events (participants affected / at risk) | 13/17 | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A, Treatment Arm (N=17) | B, Control Arm (N=10)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A, Treatment Arm (N=17) | B, Control Arm (N=10)
Constipation (Gastrointestinal disorders) | 9 (9) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Infrequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must in advance inform and provide to the sponsor a copy of the proposed publication. The sponsor may request that the PI remove confidential information from the publication.

DOCUMENTS (2):
  • Study Protocol (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT05258773/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT05258773/SAP_001.pdf